CLINICAL TRIAL: NCT03263312
Title: Multimodality Biomarkers for Noninvasive Assessment of the Fontan Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maria Bano (Other)
Responsible Party: Sponsor-Investigator, Maria Bano, Assistant Professor, Children's Medical Center Dallas
Organization: Children's Medical Center Dallas (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122016-037
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Single-ventricle; Myocardial Fibrosis
Keywords: myocardial fibrosis; exercise training; Fontan
MeSH Terms: conditions — Univentricular Heart | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fontan Patients (Experimental): All Fontan patients included in this study will be part of an exercise intervention 2-6 times/week for 3-6 months.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Exercise training all patients enrolled.
  Other Names: Training

SUMMARY:
This is a single center prospective longitudinal exercise training study and will enroll approximately 50 Fontan patients and 20 controls of a similar age, gender, BMI and physical activity level between the ages of 10-40 years.

Participants will undergo an MRI of the Fontan circulation. This will include imaging of the heart, lung and liver. This will include specific imaging for tissue characterization and assessment of myocardial fibrosis, liver fibrosis and disproportionate pulmonary blood flow. The investigators will then draw blood (approximately 10 ml) for assessment of serum biomarkers and circulating microRNAs of interest. The participants will undergo exercise testing and will then start a 3-6 month long cardiac rehabilitation program. After the 3-6 month study period the participants will return back for a follow up and repeat all the testing completed at enrollement.

DETAILED DESCRIPTION:
This is a single center prospective longitudinal study and will enroll approximately 50 Fontan patients and 20 controls of a similar age, gender, BMI and physical activity level between the ages of 10-40 years. The investigators will enroll from pediatric cardiology and heart failure clinics and inpatient care units at Children's Health Dallas, adult congenital heart disease clinics and inpatient care units at Clements University Hospital and the Clinical Heart Center. This study will evaluate the multimodality biomarkers for assessment of Fontan circulation including heart, liver and lung and change in these markers with exercise training.

Participants will receive an MRI of the Fontan circulation. This will include imaging of the heart, lung and liver. A blood draw (approximately 10 ml) for assessment of serum biomarkers and circulating microRNAs of interest will be completed. The participants will also complete exercise testing and will then start a 3-6 month long cardiac rehabilitation program. Frequent phone follow up (conducted by the research staff) and regular download of data from heart rate monitors will ensure adherence.

After the 3-6 month study period the participants will return for a follow up and repeat all testing completed at enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a congenital heart defect that leads to single ventricle physiology
* Previously performed TCPA surgery
* Current age 10 years to 40 years
* Informed consent

Exclusion Criteria:

* History of exercise intolerance (peak VO2<12ml/kg/min)
* Unstable arrhythmia at the time of screening
* Listed or being evaluated for heart transplantation
* Pregnancy or breast feeding
* Patient with pacemaker, AV block other than 1st degree block, sick sinus syndrome or other arrhythmia that may influence ability to perform exercise test or magnetic resonance imaging

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | 6 months
  Improvement in Peak VO2 with 6 months of exercise training

CONTACTS AND LOCATIONS:
Locations (1):
- Children'sMCD, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bano M, Hussain T, Samels MR, Butts RJ, Kirk R, Levine BD. Cardiovascular remodelling in response to exercise training in patients after the Fontan procedure: a pilot study. Cardiol Young. 2024 Mar;34(3):604-613. doi: 10.1017/S1047951123003153. Epub 2023 Sep 4. PMID 37664999